CLINICAL TRIAL: NCT06287671
Title: Colorectal OmiCs and Oncofetal Chondroitin Sulfate-modified Proteoglycans
Brief Title: Colorectal Omics and OfCS Proteoglycans
Acronym: COCO
Status: Recruiting | Type: Observational
Sponsor: Claus Anders Bertelsen, PhD, MD (Other)
Collaborators: Viborg Regional Hospital (Other)
Responsible Party: Sponsor-Investigator, Claus Anders Bertelsen, PhD, MD, Clinical research professor, consultant colorectal surgeon, Nordsjaellands Hospital
Organization: Nordsjaellands Hospital (Other)
Other Study IDs: COCO
Record Dates: First submitted 2024-02-22; First posted 2024-03-01 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Colorectal Cancer; Diverticulitis, Colonic; Inflammatory Bowel Diseases; Stoma Colostomy
MeSH Terms: conditions — Colorectal Neoplasms; Diverticulitis, Colonic; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood plasma Tumor tissue from participants with colorectal cancer
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study cohort: Patients undergoing elective colorectal resection or stoma closure
  Interventions: Procedure: Colorectal resection or stoma closure

INTERVENTIONS:
Procedure: Colorectal resection or stoma closure — Elective open or minimally invasive resection for colorectal cancer, IBD or other benign colorectal disorder, or stoma closure

SUMMARY:
This observational study aims to test proteomics, metabolomics and proteoglycans as predictors of postoperative complications after colorectal surgery and as biomarkers of colorectal cancer.

The main questions to answer are:

* can these biomarkers predict anastomotic leakages
* can these biomarkers predict recurrence after colorectal cancer
* can these biomarkers be used as diagnostic tests for colorectal cancer
* can these biomarkers be identified in the tumor

Participants will undergo elective colorectal resection or stoma closure.

DETAILED DESCRIPTION:
The prospective cohort study will include 1,000 patients undergoing elective colorectal resections or colostomy reversal at two colorectal centers in Denmark. Repeating study blood samples will be collected on each postoperative day (POD) 1-4 or until discharge. If the participants are diagnosed with cancer, blood sampling is planned 26-35 days after the index procedure, and after one, two, and three years, a tumor biopsy will be taken from the fresh specimen in the operation theatre.

Analyses of blood plasma and tissue for oncofetal chondroitin sulfate (ofCS) proteoglycans, proteomics, and metabolomics will be performed on those repeating blood samplings to:

* To investigate whether metabolomics, proteomics, and ofCS techniques can identify new biomarkers where charges in plasma levels can predict or detect subclinical AL (primary outcome) and other major postoperative complications after colorectal surgery and prediction of 90-day and three-year mortality.
* To investigate whether the APOE genotype is associated with the risk of AL and other major postoperative complications and long-term outcomes, i.e., recurrence and mortality, after colorectal surgery.
* To examine whether metabolomics and proteomics can identify new biomarkers predicting recurrence after colorectal cancer resections.
* To identify other potential biomarkers that might enable early cancer diagnosis.
* Whether proteoglycans can be used as a diagnostic test with a high degree of separability to identify tumor markers that are usable in a clinical setting (primary outcome). Participants with colorectal cancer will be compared with a control group of participants with benign conditions.
* Whether the level of proteoglycans measured correlates to the tumor load.
* Whether the proteoglycans and proteomics detected in plasma are presented in tumor tissue from the resected specimen.
* Whether the proteoglycans detected can be used as tumor markers with a high degree or measure of separability for monitoring recurrence after colorectal cancer in a clinical setting (primary outcome).

Postoperative and follow-up data will be collected prospectively for the electronic health records.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed or with suspicion of colorectal cancer or adenoma, inflammatory bowel disease, late complications to colon diverticulosis, colostomy reversal or other diagnoses requiring colorectal resection.
* Patients planned to undergo elective surgical procedures coded as KJFB20-KJFB99, KJFG30-37 or KJGB00-97 according to the Danish modification of the NOMESCO Classification of Surgical Procedures
* Able to speak Danish, English, or other languages where professional interpretation is available
* Able to give informed consent

Exclusion Criteria:

* Patients undergoing synchronous: liver resection (patients undergoing metastasectomies can be included); total gastrectomy or cardia resection; Whipple's procedure or another major pancreatic resection (resections of the pancreatic tail can be included); total or partial nephrectomies or cystectomy
* Patients previously included in the study
* Patients known to be pregnant (pregnancy test not required)
* Non-resident in Denmark

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients planned for elective colorectal surgery
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-10-08 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of anastomotic leakage diagnosed by CT-scan or reoperation | 30 days
  Anastomotic leakage after colorectal resection with anastomosis or stoma closure
Rate of major postoperative complications | 30 days
  Major postoperative complication (Clavien-Dindo score 3B or higher, and DVT and pulmonary embolism) after colorectal resection with anastomosis or stoma closure
Short-term mortality | 90 days
  Postoperative mortality after colorectal resection with anastomosis or stoma closure
Recurrence after colorectal cancer | 4 years
  Recurrence after radical resection, diagnosed by imaging modalities or tissue biopsy
Diagnostic value of omics and other biomarkers detecting colorectal cancer | 30 days
  Identifying omics and chondroitin sulfate-modified proteoglycans that can be used i a clinical setting to identify colorectal cancer patients
Correlation between biomarker in plasma and tissue | 30 days
  Does presence of tumor markers in blood plasma correlate with the same tumor makers in the tumor tissue

CONTACTS AND LOCATIONS:
Overall Officials: Claus A Bertelsen, PhD, Study Chair — Department of Surgery, Copenhagen University Hospital - North Zealand
Locations (2):
- Denmark (2):
  - Nordsjaellands Hospital, Hillerød
  - Regionshospitalet Viborg, Viborg

IPD SHARING:
Plan to Share IPD: No
Results will be published by the investigators in academic journals. Sharing of generated study data will be carried out in several different ways. After acceptance from the participant and the ethics committee of the Capital Region of Denmark, individual participant data and blood plasma will be available to potential collaborators interested in colorectal disorders.